CLINICAL TRIAL: NCT03680846
Title: A Multi-Center, Prospective, Pragmatic, Randomized, Controlled Clinical Trial to Compare HF10 Therapy to Conventional Medical Management in the Treatment of Non-Surgical Refractory Back Pain
Brief Title: Comparison of HF10 Therapy Combined With CMM to CMM Alone in the Treatment of Non-Surgical Refractory Back Pain
Acronym: NSRBP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Nevro Corp (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA2018-2 US NSRBP
Record Dates: First submitted 2017-11-14; First posted 2018-09-21 (Actual); Last update posted 2021-10-12 (Actual); Status verified 2021-10

CONDITIONS: Back Pain
MeSH Terms: conditions — Back Pain

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- CMM (Other): Conventional Medical Management
  Interventions: Other: CMM
- HF10 + CMM (Active Comparator): Addition of HF10 therapy to CMM
  Interventions: Device: HF10 Therapy; Other: CMM

INTERVENTIONS:
Device: HF10 Therapy — Senza 10 kHz Spinal Cord Stimulation
  Arms: HF10 + CMM
Other: CMM — Conventional Medical Management

SUMMARY:
This study is being conducted to document the safety, clinical effectiveness and cost-effectiveness of high-frequency SCS at 10 kHz (HF10™ Therapy) delivered through the Senza system in subjects with chronic refractory back pain (with or without leg pain) who are not considered candidates for spine surgery. This study is a multi-center, prospective, randomized study to compare the two treatment groups.

ELIGIBILITY:
Key Inclusion Criteria:

1. Have been diagnosed with chronic, refractory axial low back pain with a neuropathic component and are not eligible for spine surgery
2. Have not had any surgery for back or leg pain, or any surgery resulting in back or leg pain
3. Qualifying pain score
4. Be on stable pain medications, as determined by the Investigator
5. Be willing and capable of giving informed consent
6. Be willing and able to comply with study-related requirements, procedures, and visits
7. Be capable of subjective evaluation, able to read and understand written questionnaires in the local language and are able to read, understand and sign the written inform consent

Key Exclusion Criteria:

1. Have a diagnosed back condition with inflammatory causes of back pain, serious spinal pathology and/or neurological disorders
2. Have a medical condition or pain in other area(s), not intended to be treated in this study
3. Any diagnosis or known condition that can impact reporting of study outcomes as determined by the Investigator
4. Be benefitting within 30 days prior to enrollment from an interventional procedure to treat back and/or leg pain
5. Have any addictions as determined by the Investigator
6. Have an existing drug pump and/or SCS system or another active implantable device such as a pacemaker
7. Have prior experience with neuromodulation devices
8. Other general exclusions applicable for SCS devices
9. Be involved in an injury claim under current litigation
10. Have a pending or approved worker's compensation claim

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 211 (Actual)
Dates: Start 2018-09-05 (Actual); Primary Completion 2020-10-06 (Actual); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Difference between treatment groups in responder rates. | 3 Months
  Responder is defined as a subject who has at least 50% reduction in pain from Baseline as assessed by a 10 cm Visual Analog Scale (VAS)

SECONDARY OUTCOMES:
Change in Disability as Measured by Oswestry Disability Index | 6 months
  Percentage of subjects with at least 10 point decrease from Baseline in Oswestry Disability Index (ODI) score
Percentage change from baseline in back pain intensity (as assessed by VAS) | 6 months
Changes in Quality of Life (QOL) as measured by EuroQol EQ-5D-5L questionnaire | 6 months
  It measures the subject's health state as assessed in 5 dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) each with 5 levels. In addition there is an EQ VAS which records the patient's self-rated health on a vertical visual analogue scale. The scores on these five dimensions can be presented as a health profile or can be converted to a single number summary called the "index value".
Global impression of change | 6 months
  Proportion of subjects reporting "better" or "great deal better" on the Patient Global Impression of Change (PGIC) questionnaire
Change from baseline in opioid equivalent medication usage in each group | 6 months
Neurological assessment | 3, 6 and 12 months
  Assessment of motor, sensory and reflex functions. Clinicians shall characterize the findings as improved, maintained, or a deficit as compared with baseline status.
Incidences of adverse events | 3, 6 and 12 months

OTHER OUTCOMES:
Observational Outcomes on reduction in pain using a 10 cm Visual Analog Scale (VAS) | 24 months
  Percentage change in back pain
Observational Outcomes on disability using Oswestry Disability Index scores | 24 months
  Percentage change from Baseline in ODI score
Observational Outcomes on Health related quality of life evaluation as measured by the 5 dimension EuroQol EQ-5D-5L questionnaire | 24 months
  Change in quality of life index compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: David Caraway, MD, Study Director — Nevro Corp
Locations (1):
- Nevro Corp, Redwood City, California, United States

REFERENCES:
- [Derived] O'Connell NE, Ferraro MC, Gibson W, Rice AS, Vase L, Coyle D, Eccleston C. Implanted spinal neuromodulation interventions for chronic pain in adults. Cochrane Database Syst Rev. 2021 Dec 2;12(12):CD013756. doi: 10.1002/14651858.CD013756.pub2. PMID 34854473
- [Derived] Patel N, Calodney A, Kapural L, Province-Azalde R, Lad SP, Pilitsis J, Wu C, Cherry T, Subbaroyan J, Gliner B, Caraway D. High-Frequency Spinal Cord Stimulation at 10 kHz for the Treatment of Nonsurgical Refractory Back Pain: Design of a Pragmatic, Multicenter, Randomized Controlled Trial. Pain Pract. 2021 Feb;21(2):171-183. doi: 10.1111/papr.12945. Epub 2020 Sep 26. PMID 33463027